CLINICAL TRIAL: NCT07178366
Title: Impact of Double Plasma Separation and Adsorption on Patients With Acute on Chronic Liver Failure- A Prospective Open-label Randomized Controlled Trial
Brief Title: Double Plasma Separation and Adsorption in Acute-on-Chronic Liver Failure (DPMAS-ACLF Trial)
Acronym: DPMAS-ACLF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Rakhi Maiwall, Professor of hepatology, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2025/117/MA01; IEC Approval Number (Other: Institute of Liver and Biliary Sciences (ILBS))
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Acute-on-Chronic Liver Failure (ACLF)
Keywords: ACLF; DPMAS; Lactate; Sepsis; Liver support
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Sepsis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio into two parallel groups. One group will receive standard medical therapy (SMT) alone, while the other group will receive SMT plus Double Plasma Molecular Adsorption System (DPMAS). Randomization will be open-label, and each participant will remain in the assigned group for the duration of the study.
Masking Description: This is an open-label randomized controlled trial. No masking will be performed for participants, care providers, investigators, or outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy (SMT) Group (Active Comparator): Participants will receive standard medical therapy alone, which may include nutritional support, lactulose, bowel wash, albumin, vasopressors (norepinephrine/terlipressin), antibiotics, antivirals for HBV reactivation, renal replacement therapy, and intensive care support as per institutional guidelines.
  Interventions: Other: Standard medical therapy (SMT)
- SMT + Double Plasma Molecular Adsorption System (DPMAS) (Experimental): Participants will receive standard medical therapy plus DPMAS therapy. DPMAS involves extracorporeal liver support using two sequential hemoadsorption cartridges (BS330 ion exchange resin and HA330-II neutral macroporous adsorption resin). A minimum of 2 sessions (3-4 hours each) will be given in the first 7 days, with additional sessions if partial response is observed.
  Interventions: Other: Standard medical therapy (SMT); Device: Double Plasma Molecular Adsorption System (DPMAS)

INTERVENTIONS:
Other: Standard medical therapy (SMT) — Standard medical therapy includes nutritional support (25-30 kcal/kg/day), lactulose, bowel wash, albumin, vasopressors (norepinephrine/terlipressin), antibiotics, antivirals for HBV reactivation, renal replacement therapy, and intensive care support as per institutional guidelines.
Device: Double Plasma Molecular Adsorption System (DPMAS) — DPMAS therapy uses extracorporeal liver support with two sequential hemoadsorption cartridges (BS330 ion exchange resin and HA330-II neutral macroporous adsorption resin). Minimum 2 sessions (3-4 hours each) are performed within the first 7 days, with additional sessions if partial response is observed.
  Arms: SMT + Double Plasma Molecular Adsorption System (DPMAS)

SUMMARY:
Acute-on-chronic liver failure (ACLF) is a serious condition in which patients with chronic liver disease suddenly develop severe liver injury, leading to inflammation, organ failure, and very high short-term mortality. Standard medical treatment can help, but many patients still do poorly without liver transplantation.

This study will test whether Double Plasma Molecular Adsorption System (DPMAS), an extracorporeal blood purification therapy, can improve outcomes in ACLF patients. DPMAS works by filtering the blood through special adsorption columns that remove harmful substances such as bile acids, toxins, and inflammatory molecules.

In this randomized controlled trial, adult patients with ACLF will be randomly assigned to receive either:

Standard medical therapy alone, or

Standard medical therapy plus DPMAS.

The main goal is to see whether DPMAS can improve liver function and reduce disease severity within 14 days. Other outcomes include survival without liver transplant at 28 days, improvement in organ functions, reduction in inflammation, and safety of the procedure.

The study will be conducted at the Institute of Liver and Biliary Sciences (ILBS), New Delhi, India, and will enroll about 56 participants over one year.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) is characterized by acute deterioration of liver function in patients with chronic liver disease, leading to systemic inflammation, organ failure, and high short-term mortality. Current treatment is largely supportive, and liver transplantation is often the only curative option, but many patients are not eligible or die while awaiting transplant.

Recent evidence suggests that systemic inflammation, bile acid accumulation, and damage-associated molecular patterns (DAMPs) play key roles in the progression of ACLF. Extracorporeal liver support systems such as plasma exchange have shown benefit in selected patients by reducing inflammation and improving short-term survival.

The Double Plasma Molecular Adsorption System (DPMAS) is a novel extracorporeal therapy that combines plasma separation with sequential adsorption columns. These columns are designed to remove bile acids, bilirubin, cytokines, and other toxins from the circulation. Early studies suggest that DPMAS may improve organ function and reduce mortality in ACLF.

This prospective, open-label, randomized controlled trial will compare standard medical therapy (SMT) alone versus SMT plus DPMAS in adult patients with ACLF (AARC grade II or higher). The primary outcome is an improvement in AARC grade by 1 at day 14 (7 days off treatment). Secondary outcomes include transplant-free survival at 28 days, changes in systemic inflammation, renal and hemodynamic function, bilirubin and bile acid levels, development of infections or new organ failures, and safety of the therapy.

A total of 56 participants will be enrolled and randomized equally into the two study groups. Patients in the intervention arm will undergo a minimum of two DPMAS sessions within the first seven days, with additional sessions as clinically indicated. Participants will be followed for up to 90 days for survival and clinical outcomes.

The study is investigator-initiated and conducted at the Institute of Liver and Biliary Sciences (ILBS), New Delhi, India. Ethical approval has been obtained from the ILBS Institutional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* ACLF patients of any etiology with systemic inflammatory response syndrome and AARC grade II or more.

Exclusion Criteria:

* Patients eligible for corticosteroids for severe alcohol-associated hepatitis related ACLF (other than hydrocortisone according to Surviving Sepsis Campaign Guidelines 2021 which is 50 mg iv q 6 h for management of refractory shock
* Hepatocellular carcinoma or any extrahepatic malignancy,
* Active fungal sepsis
* Disseminated intravascular coagulation
* Hemodynamic instability requiring norepinephrine >0.20ug/kg/min
* Patients with coma of non-hepatic origin
* Patients with PaO2/FiO2 ratio <150
* Pregnancy
* Comorbidities associated with poor outcomes (severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease, chronic kidney disease) and patients with post-resection liver failure
* Patients with fibrinogen <110 and/or platelets less than 50,000
* Patients with oliguria with urine output less than 400 ml/day
* Lack of informed consent
* Patient enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in AARC ACLF grade by one at day 14 (after 7 days off treatment) | 14 days
  Proportion of participants who show an improvement of at least one grade in the Asian Pacific Association for the Study of the Liver acute-on-chronic liver failure (AARC ACLF) score at day 14, assessed after a treatment-free interval of 7 days from randomisation.

SECONDARY OUTCOMES:
Transplant-free survival | 28 Days
  Proportion of participants alive without liver transplantation at 28 days after randomization.
Change in cytokine levels | 14 days
  Change in serum cytokine concentrations (IL-6, TNF-α, IL-10) measured by multiplex bead-based immunoassay (e.g., Luminex platform) from baseline to Day 14
Change in DAMPs | 14 days
  Change in circulating damage-associated molecular patterns (HMGB1 and mitochondrial DNA) measured by ELISA and quantitative PCR, respectively, from baseline to Day 14
Change in serum bilirubin levels | 14 days
  Change in serum bilirubin concentration from baseline to Day 14.
Change in serum bile acid levels | 14 days
  Change in serum bile acid concentration from baseline to Day 14.
Change in serum creatinine levels | 14 days
  Change in serum creatinine concentration from baseline to Day 14.
Change in urine output | 14 days
  Change in urine output from baseline to Day 14
Change in mean arterial pressure | 14 days
  Change in mean arterial pressure from baseline to Day 14
Change in vasopressor requirement | 14 days
  Change in vasopressor requirement from baseline to Day 14
Incidence of new infections | 28 days
  Number of participants who develop new infections during the follow-up period
Development of new organ failures | 28 days
  Proportion of participants with new organ failures, assessed using the CLIF-OF score.
Safety and tolerability of DPMAS | Upto 90 days
  Incidence of adverse events such as hypotension, bleeding, sepsis, metabolic disturbances, or allergic reactions during therapy and follow-up.